CLINICAL TRIAL: NCT06940297
Title: DART: Phase II Study of Dasatinib and Quercetin in Patients With Relapsed, Refractory Multiple Myeloma Receiving CAR-T Therapy
Brief Title: Dasatinib and Quercetin With CAR-T Therapy for the Treatment of Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240801; NCI-2025-02490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-002915 (Other: Mayo Clinic Institutional Review Board); MC240801 (Other: Mayo Clinic); P50CA186781 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Biopsy; Specimen Handling; bis(3-bis(4-chlorophenyl)methyl-4-dimethylaminophenyl)amine; Cyclophosphamide; Dasatinib; fludarabine; Magnetic Resonance Spectroscopy; Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Dasatinib, quercetin, chemotherapy, CAR-T) (Experimental): Patients receive dasatinib by mouth (PO) once a day (QD) and quercetin PO twice a day (BID) on days -7 and -6 and cyclophosphamide IV over 60 minutes and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity. Patients then receive CAR-T IV on day 0. Patients receive dasatinib PO QD and quercetin PO BID on days 28, 29, 58, 59, 88 and 89 in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and/or PET, tumor biopsy, bone marrow aspirate and biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Biological: Ciltacabtagene Autoleucel; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Dasatinib; Drug: Fludarabine; Procedure: Positron Emission Tomography; Drug: Quercetin

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Biological: Ciltacabtagene Autoleucel — Given IV
  Other Names: Autologous Anti-B-cell maturation antigen (BCMA) CAR-T Cells JNJ-68284528; Autologous Bi-epitope BCMA-targeted CAR T-cells JNJ-68284528; Autologous Bi-epitope CAR T-cells JNJ-68284528; CARVYKTI; Cilta-cel; JNJ 68284528; JNJ-68284528; JNJ68284528; LCAR B38M; LCAR-B38M; LCAR-B38M-transduced CAR-T Cells JNJ-68284528; LCARB38M; Autologous Anti-BCMA CAR-T Cells JNJ-68284528
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Quercetin — Given PO
  Other Names: 2-(3,4-dihydroxyphenyl)-3,5,7-trihydroxy-4H-1-benzopyran-4-one; 2-(3,4-dihydroxyphenyl)-3,5,7-trihydroxy-chromen-4-one; C.I. Natural Yellow 10

SUMMARY:
This phase II trial tests how well giving dasatinib and quercetin with cyclophosphamide, fludarabine and chimeric antigen receptor (CAR)-T cell therapy works in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Dasatinib is in a class of medications called tyrosine kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply, which may help keep cancer cells from growing. Quercetin is a compound found in plants that may prevent multiple myeloma from forming. Chemotherapy such as cyclophosphamide and fludarabine are given to help kill any remaining cancer cells in the body and to prepare the bone marrow for CAR-T therapy. Chimeric antigen receptor T-cell Therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Giving dasatinib and quercetin with cyclophosphamide, fludarabine and CAR-T cell therapy may kill more cancer cells in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Relapsed or refractory multiple myeloma who has had at least 3 prior lines of therapies including a proteasome inhibitor, immunomodulatory drug (IMiD) and anti-CD38 monoclonal antibody (mAb)
* Ciltacabtagene autoleucel (Carvykti) available for patient
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 8.0 g/dL (obtained ≤ 14 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3 (obtained ≤ 14 days prior to registration)
* Platelet count ≥ 50,000/mm^3 (obtained ≤ 14 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 14 days prior to registration)

  * Note: Patients with Gilbert's syndrome must have a total bilirubin of ≤ 3 x ULN (obtained ≤ 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2 x ULN (obtained ≤ 14 days prior to registration)
* Alkaline phosphatase ≤ 1.5 x ULN (obtained ≤ 14 days prior to registration)
* Calculated creatinine clearance ≥ 30 ml/min using the Cockcroft-Gault formula (obtained ≤ 14 days prior to registration)
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only

  * Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Sexually active patients and their partners must use an effective method of contraception associated with a low failure rate prior to study entry and for the duration of study participation and for at least 30 days after the last dose of study drug
* Provide written informed consent
* Willingness to provide mandatory blood and bone marrow specimens for correlative research
* Willingness to provide mandatory bone marrow cores and/or tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, or AL amyloidosis
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment.

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 1 month since completion of prior treatment
* Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential (and persons able to father a child) who are unwilling to employ adequate contraception
* Major surgery ≤ 28 days prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be HIV positive.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, or those currently receiving antiretroviral therapy with good control of HIV, are eligible for this trial
* Evidence of cardiovascular disease risk, as defined by any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of screening.
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system
  * Uncontrolled hypertension
  * History of life-threatening ventricular arrhythmias
  * QTC interval [electrocardiogram (ECG)] ≥ 450 msec
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Any medical condition that would make participation unduly hazardous
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Live vaccine ≤ 6 weeks prior to registration
* Has taken a strong inhibitor or inducer of CYP3A4/5, including grapefruit, St. John's Wort or related products ≤ 14 days prior to registration.

  * Note: If required, patients may receive a short course of strong inhibitors or inducers for treatment of symptoms, but dasatinib dose must be adjusted as indicated
* Known hypersensitivity or allergy to dasatinib or quercetin
* Patients on therapeutic doses of anticoagulants (e.g. warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc).
* On antiplatelet agents (e.g. full dose aspirin, clopidogrel etc.)

  * NOTE: Baby aspirin, if necessary for cardioprotection, will be allowed
* On quinolone antibiotic therapy for treatment or for prevention of infections products ≤10 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2031-08-15 (Estimated); Study Completion 2031-08-15 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negativity rate | At 3 months
  Defined as the number of patients who are able to achieve undetectable MRD based on bone marrow (BM) and positron emission tomography (PET) evaluations.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Assessed by the number of patients who achieve any response (partial response or better) to therapy.
Depth of response | Up to 2 years
  Assessed by the number of patients who are able to achieve different levels of response, such as partial response (PR), very good partial response (VGPR), and complete response (CR), or stringent complete response (sCR).
Progression free survival (PFS) | Up to 2 years
  Defined as the time from study registration to the time of documented disease progression or death due to any cause.
Duration of response | Up to 2 years
  Defined as the time from first documented response to the time of progression and/or death due to any cause.
Incidence of adverse events (AEs) | Up to 2 years
  AEs will be summarized per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5, and where toxicities will be defined as adverse events that are deemed to be at least possibly treatment-related. The maximum grade for each type of treatment-related AE will be recorded for each patient, and the frequency of each will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lin, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials